CLINICAL TRIAL: NCT00156520
Title: Jeanne Grace; Head Research Subjects Review Board
Brief Title: Platelet Function And Aggregometry In Patients With Aortic Valve Stenosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 10504
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-04

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — Aminocaproic Acid

INTERVENTIONS:
Drug: aprotonin; epsilon aminocaproic acid

SUMMARY:
It is known that patients with aortic stenosis, including those undergoing cardiac surgery for this problem, are prone to developing bleeding problems, particularly of the gastrointestinal tract. It is believed that the shear stress associated with blood flow through the abnormal aortic valve results in abnormal hemostasis. Abnormalities include increased proteolysis of the von Willebrand factor (vWF) and increased binding of the high molecular weight multimers of vWF to platelet membranes with subsequent inappropriate platelet aggregation. Thus, appropriate aggregation of circulating platelets is impaired. Cardiac surgery is associated with significant alterations in hemostasis. Patients undergoing cardiac surgery consume a significant percent of available blood products throughout the United States and are subjected to various and numerous risks associated with blood product transfusion. In addition, excessive postoperative bleeding is a common cause for the need to surgically re-explore the chest cavity in patients who have just undergone cardiac surgical procedures. Such additional surgery carries further cost and risk. Following surgical correction of aortic valve stenotic pathology, associated vWF abnormalities appear to reverse. However, this process can take several days. Although all cardiac surgical patients are at risk for postoperative bleeding, patients undergoing aortic valve surgery for aortic stenosis may be particularly at risk for this postoperative complication. In addition, patients with aortic valve stenosis who undergo noncardiac surgery may have a predisposition to bleeding because of similar underlying shear stress induced abnormal vWF and platelet function. The proposed study is a trial to evaluate the effectiveness of 2 different antifibrinolytic drugs in ameliorating the hemostatic defect associated with aortic stenosis. Aprotonin, an antifibrinolytic agent which also has platelet preserving actions4, will be compared to the currently used anti-fibrinolytic, epsilon aminocaproic acid (EACA).

DETAILED DESCRIPTION:
Study subjects will be competent adult patients who are scheduled to undergo elective aortic valve surgery for severe aortic stenosis. The process of informed consent will begin prior to the day of surgery either during a patient's preoperative surgery clinic visit with one of the cardiac surgeons for any patient having such a clinic visit or during the preoperative anesthesia evaluation prior to the day of surgery. At one or both of these times patients will be told of the study and given a copy of the informed consent for their reading. An opportunity for them to discuss the study at this time will be offered. Written informed consent will be obtained on the day of surgery, prior to surgery. Patients must not also require coronary artery surgery or be taking or receiving drugs that alter platelet function, including aspirin (within the past 2 weeks) or any of the modern a ADP receptor antagonists such as Plavix. As per current patient care guidelines at Strong Memorial Hospital, patients undergoing first-time single valve, non-coronary artery surgical procedures will be randomized to receive either epsilon aminocaproic acid (EACA) or aprotonin intravenously. It is anticipated that 1-3 patients will be initially enrolled as pilot subjects to get the study going smoothly and that 1-3 patients may not be completed or that their testing and/or data may be inadequate. Therefore, although the analysis will only use 40 subjects the protocol seeks permission to enroll a maximum of 24 subjects per group for a total of 48 patients.

The tests to be performed are:

1. the PFA-100, a platelet related hemostasis test which is a high shear system test of platelet function
2. the von Willebrand antigen test, an immunoassay
3. factor VIII coagulant activity test.
4. Ristocetin cofactor activity test.
5. thromboelastography (TEG), a point-of-care test of hemostatic function which includes a measure of platelet function.

(Reference ranges / coefficient of variation / SD's / for the tests are as follows:

vWF-Ag: 50 - 160% normal activity / 2 - 5% / ~5%

FVIII: 50 - 200% of normal / 4 - 7% / ~5%

Ristocetin cofactor: 60-200% of normal / ~15% / ~10%

PFA100 closure time: epinephrine <181 seconds and ADP <112 seconds / ~12% / 20 secs)

Total blood volume required from each patient for the purposes of doing the research related tests will be approximately 30 mls (1 fluid ounces or 2 tablespoons). 10 mls will be drawn from each patient's arterial line, which is routinely placed for cardiac anesthesia & surgery care, at the following time points in their care:

1. prior to induction of anesthesia
2. 5 minutes after the loading dose of either EACA or aprotonin has been administered and prior to the administration of any heparin
3. 15 minutes after the administration of protamine following termination of cardiopulmonary bypass.

Thus, no additional "needle puncture" will be necessary related to the study. Each blood sample of 10 ml will be divided into one "blue-top" (citrated) tube (3 ml) and kept on ice, one "blue-top" (citrated) tube (3 ml) and kept at room temperature, and the remainder will be used to perform the TEG.

IV. Data Analysis and Monitoring:

Statistical analysis will be performed using either a 2-sample t-test or the Mann-Whitney Test, as appropriate, to compare the two patient groups at each of the three time points. A p-value of less than 0.05 will be considered significant. All tests will be two-sided.

With a proposed sample size of N = 20 for each of the two groups, the study will have at least 80% power to yield a statistically significant result.

V. Data Storage and Confidentiality:

Data will be produced within the SMH hematology lab and then stored both on paper and on the computer in the Department of Anesthesiology and backed up on the network drive.

The principal investigator will maintain the information in a password protected file on the computer in his (their) private office.

ELIGIBILITY:
Inclusion Criteria:Study subjects will be competent adult patients who are scheduled to undergo elective aortic valve surgery for severe aortic stenosis.

- Exclusion Criteria: Potential study subjects will be excluded if they are scheduled to undergo elective aortic valve surgery for severe aortic stenosis and any other surgery simultaneously or have been taking aspirin within 6 days of surgery.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-03; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
1. the PFA-100, a platelet related hemostasis test which is a high shear system test of platelet function
  PFA-100, a platelet related hemostasis test
2. the von Willebrand antigen test, an immunoassay
  von Willebrand antigen test
3. factor VIII coagulant activity test.
  Factor VIII coagulant activity test
4. Ristocetin cofactor activity test.
5. thromboelastography (TEG), a point-of-care test of hemostatic function which includes a measure of platelet function.

SECONDARY OUTCOMES:
thromboelastography
  thromboelastography point of care test of hemostatic function

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Bailey, MD', Principal Investigator — University of Rochester, Rochester, NY 14642
Locations (1):
- Strong Memorial Hospital, University of Rochester, Rochester, New York, United States